CLINICAL TRIAL: NCT02373917
Title: Characterization of Methylation Patterns in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Lung-RND-001
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Blood samples
  2. Sputum samples
  3. saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: patient who in the biopsy showed lung cancer
- control group: patient who in the biopsy showed not to have lung cancer

SUMMARY:
In this study the investigators will collect Blood,sputum and saliva samples for Characterization of Methylation Patterns in lung Cancer.

DETAILED DESCRIPTION:
Lots of information about the relationship between changes in methylation patterns and various diseases are accumulated in recent years. Characterization of methylation changes that occur in cancer may contribute to the development of methods for early detection of cancer by detecting cancer cells in liquids. Early detection of such changes and their correlation examining different cancers may lead to a diagnostic tool for the early detection of cancers and improve the treatment of these patients. Detection by molecular analysis can be a sensitive method and non-invasive early diagnosis of the disease In this study the investigators will collect Blood,sputum and saliva samples for Characterization of Methylation Patterns in lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected lung tumor

Exclusion Criteria:

* Patients who have active disease other than lung cancer during the sample collecting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who come to the medical center for the diagnosis of lung cancer.
Sampling Method: Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Characterization of Methylation Patterns in lung Cancer | two years
  Collecting and analyzing samples

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Ganor, MD, Study Director — Nucleix Ltd.
Locations (1):
- Sha'are Tzedaek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Gaga M, Chorostowska-Wynimko J, Horvath I, Tammemagi MC, Shitrit D, Eisenberg VH, Liang H, Stav D, Levy Faber D, Jansen M, Raviv Y, Panagoulias V, Rudzinski P, Izbicki G, Ronen O, Goldhaber A, Moalem R, Arber N, Haas I, Zhou Q. Validation of Lung EpiCheck, a novel methylation-based blood assay, for the detection of lung cancer in European and Chinese high-risk individuals. Eur Respir J. 2021 Jan 14;57(1):2002682. doi: 10.1183/13993003.02682-2020. Print 2021 Jan. PMID 33122336